CLINICAL TRIAL: NCT05202886
Title: "LiverColor": AN ALGORITHM QUANTIFICATION OF LIVER GRAFT STEATOSIS USING MACHINE LEARNING AND COLOR IMAGE PROCESSING
Brief Title: "LiverColor": Machine Learning in Liver Photographs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Vall d'Hebron (Other)
Responsible Party: Principal Investigator, Concepción Gomez Gavara, PhD, Hospital Vall d'Hebron
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PR(AG)04/2018
Record Dates: First submitted 2021-06-08; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Brain Death; Liver Steatosis
Keywords: machine learning; liver donor (DBD); liver steatosis; liver pictures; liver pool
MeSH Terms: conditions — Brain Death; Fatty Liver

STUDY DESIGN:
Intervention Model Description: Liver from deceased donors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver from deceased donors (Experimental): This study included all consecutive subjects with chronic liver disease who underwent LT for the first time with a deceased donor liver
  Interventions: Diagnostic Test: Liver from deceased donors

INTERVENTIONS:
Diagnostic Test: Liver from deceased donors — Liver donors photographed

SUMMARY:
The main goal of this project is to create a machine learning model in order to quantify liver steatosis in liver donor faster, more objective and reliable than histological analysis and surgeons point-of-view.

DETAILED DESCRIPTION:
Surgeons (junior and senior operators) from the HBP & Transplantation Unit took the pictures. They were taken after the laparotomy and before any type of surgical procedure. For each deceased donor case, a total of 5 pictures were taken: one for the left lobe and another for the right one before undergoing a surgical biopsy, two more (one for the left and one for the right lobe) after the histological analysis, near to the site of the surgical biopsy, and finally, one picture after liver perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Livers from donor donor brain death with informed consent before inclusion in the study was obtained from all participants or families.

Exclusion Criteria:

* Age < 18 years old
* Donor after cardiac death
* Split
* Cholestasis due to a biliary obstruction
* Total bilirubin levels above 2,5 mg/dL
* Glutamic oxaloacetic transaminase (SGOT)/ serum glutamatepyruvate transaminase (SGPT) levels and gamma-glutamyl transaminase (GGT) levels above 400 U/L
* Cirrhotic livers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2018-06-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The main goal of this project is to create a machine learning model in order to quantify liver steatosis in liver donor faster, more objective and reliable than histological analysis and surgeons point-of-view. | 4 weeks
  Accuracy

SECONDARY OUTCOMES:
To build an image dataset to evaluate postransplant liver function. | 1 week
  PDF will be evaluated according to Olthoff criteria

CONTACTS AND LOCATIONS:
Overall Officials: Concepcion Gómez-Gavara, PhD, Principal Investigator — Vall D´Hebron University Hospital
Locations (1):
- Concepción Gómez-Gavara, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No